CLINICAL TRIAL: NCT01854112
Title: Helical Irradiation of Total Skin (HITS) for T Cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH No. 101115-E
Record Dates: First submitted 2013-05-09; First posted 2013-05-15 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2013-05

CONDITIONS: T-cell Lymphoma
Keywords: Helical tomotherapy; total skin electron therapy; TSEB; irradiation 5.
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- T-cell lymphoma

SUMMARY:
Radiation therapy, total skin electron therapy (TSET), achieves a high response rate and is an effective treatment for cutaneous T-cell lymphoma affecting the superficial region 1. One the most widely used TSET techniques consists of six dual fields initially developed at Stanford University 2. Dosimetrically, TSET at energies of about 3-7 MeV at the surface of a standing patient may result in significant dose variations due to variable skin distance, self shielding, irradiated fields overlapping and patient motion. Deviations occur from the prescription dose up to 40% and the surface dose inhomogeneity as much as 90% in body areas such as the perineum and eyelid, are revealed in the literature. To improve this condition, a selection of patients with advanced skin disease and regional extension could be cured by a combination of TSEB and photon beam irradiation.

Helical tomotherapy (HT) has advantages in irradiating extended volumes with treatment length of up to 160 cm, continuously in a helical pattern without the need for field junction. Total marrow irradiation (TMI) via HT with low toxicities for bone marrow transplantation of Asia multiple myeloma patients could be feasible . A study of HT for total scalp irradiation has also shown that the employment of directional and complete blocking on the inner structures can effectively force the tangential delivery of the majority of beamlets to the PTV, which can limit the treatment depth.

Using HT, an image-guided intensity-modulated radiotherapy, to replace conventional TSI technique to increase dose delivery and decrease toxicities could be a workable and feasible. Here, we applied TSI via HT (HITS) for a woman with T cell lymphoma failure by chemotherapy, topic UV irradiation and local radiotherapy (RT) in MMH to overcome the surface dose inhomogeneity by conventional RT. Additionally, we will compare the advantages and disadvantages between the plan of HT and conventional RT for TSI.

DETAILED DESCRIPTION:
Helical tomotherapy planning

Patient will dress the diving suit (3 mm thick) to create bolus effect. AccuFix™ Cantilever Board™ with shoulder depression and thermoplastic fixation were used for head and shoulder immobilization. BlueBagTM immobilization system (Medical Intelligence) was used to fix main trunk and extremities. Both immobilization systems provide a consistent treatment position from the initial computed tomography (CT) scanning, pretreatment megavoltage CT (MVCT) imaging to final treatment delivery. For tomotherapy treatment planning, a CT image set of the whole body was required. The patients were scanned in a large bore (75 cm) CT scanner (Siemens, SOMATOM Definition, Dual source computed tomography system). Because most critical organs are located in the central part of the body, therefore two image sets were scanned with 2.5 mm and 5 mm for upper and lower part, respectively. The level at 15 cm above knee was used as a reference point to separate the upper and lower set. The geometric edges of both fields were abutted at the HT treatment's 50% isodose plane.

Both image sets were restored on a Pinnacle workstation using the Pinnacle Launch Pad Restore utility then using the Philips Pinnacle3 treatment planning system for contouring because the HT planning system has no such capability. After that, the plan was transferred to the Tomotherapy Hi Art Planning system (Tomotherapy, Inc., Madison, Wisconsin, USA). The clinical target volume (CTV) included the entire body surface system with subcutaneous 0.5 cm. To account for set-up variability and breathing motion, a planning target volume (PTV) was generated with a 0.5 cm margin The prescription dose was 75 cGy/fraction in 4 times/wk for total skin area and for tumor area. Total doses of 30 Gy to 95% of the PTV are delivered to the total skin area and tumor part, respectively. The normal tissue dose constraints utilized were based on the results of the survey of the clinical outcome of the target dose and dose limits to various organs at risk (OARs) such as the brain, optic chiasm, optic nerves, lenses, eyes, parotid glands, oral cavity, thyroid gland, bilateral lungs, esophagus, heart, liver, spleen, pancreases, kidneys, bowel, bladder, uterus and vagina. Maximum importance was given to target dose coverage. The constraints on dose and penalty were adjusted accordingly during optimization. The field width, pitch, and modulation factor (MF) used for the treatment planning optimization were 2.5, 0.287 cm, and 3.5, respectively. The dose volume histograms (DVHs) were calculated for the target and individual OARs. Toxicity of treatment was scored according to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0).

Image guidance:

Daily check of patient positioning was performed by the MVCT system integrated in the tomotherapy machine. Briefly, before every treatment, MVCT scans were taken in selected regions using the normal mode (4 mm slice thickness) of the body and fused with the treatment planning CT scan using bony anatomy and soft tissue images such as the lungs. Three sets of MVCT scan (scan 1, orbits to T4; scan 2, T10 to the ischial tuberosities; scan 3, 15 cm above knee to 15 cm below knee) were performed to the check the patient's whole body alignment. MVCT scans were obtained. Image fusions were evaluated by the attending physician and physicist. Any translational shifts suggested by the image fusion results were applied to the final patient setup before treatment delivery. The tolerance of setup error allowed only a 5-mm difference between the three scans in any of the three translation directions and 1° of difference in roll. Additional selected MVCT scans were performed after treatment to verify patient immobilization.

ELIGIBILITY:
Inclusion Criteria:

T-cell lymphoma

Exclusion Criteria:

-

Ages: 37 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: T-cell lymphoma
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Skin lesions size | every month from treatment up to half year